CLINICAL TRIAL: NCT04905654
Title: Migraine Inducing Effect of Levcromakalim in Patients With Migraine With Aura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Andreas Vinther Thomsen, Principal Investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-20049785
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Headache, Migraine; Aura
Keywords: Levcromakalim
MeSH Terms: conditions — Migraine Disorders; Epilepsy | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator)
  Interventions: Drug: Levcromakalim
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — To investigate the role of levcromakalim compared with placebo in migraine with aura patients
  Arms: Levcromakalim
Drug: Saline — To investigate the role of levcromakalim compared with placebo in migraine with aura patients
  Arms: Saline

SUMMARY:
To investigate the migraine inducing effect of levcromakalim in patients with migraine with aura.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with aura patients of both sexes.
* 18-70 years.
* 50-100 kg.

Exclusion Criteria:

* Headache less than 48 hours before the tests start
* Daily consumption of drugs of any kind that investigator deems might affect study results or safety.
* Pregnant or nursing women.
* Cardiovascular disease of any kind, including cerebrovascular diseases.
* Tension type headache (TTH) according to International Classification of Headache Disorders version 3 more than 5 times a month on average during the past year
* Known cluster headache according to International Classification of Headache Disorders version 3.
* Psychiatric disorder
* Smoking or abuse of drugs or alcohol
* Hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg) on day of inclusion.
* Hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg) on day of inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Headache incidence | 10 minutes before until 24 hours after infusion of levcromakalim or placebo
  Difference in incidence of headache following infusion of levcromakalim compared to placebo in patients with migraine with aura.
Migraine incidence | 10 minutes before until 24 hours after infusion of levcromakalim or placebo
  Difference in incidence of migraine-like headache following infusion of levcromakalim compared to placebo in patients with migraine with aura.
Aura incidence | 10 minutes before until 24 hours after infusion of levcromakalim or placebo
  Difference in incidence of migraine aura following infusion of levcromakalim compared to placebo in patients with migraine with aura.

SECONDARY OUTCOMES:
Headache intensity | 10 minutes before until 24 hours after infusion of levcromakalim or placebo
  The area under the curve (AUC) for headache following infusion of levcromakalim compared to placebo in patients with migraine with aura
Heart rate | 10 minutes before until 120 minutes after infusion of levcromakalim or placebo
  Change in heart rate measured in Beats per minute (BPM) following infusion of levcromakalim compared to placebo in patients with migraine with aura
Blood pressure | 10 minutes before until 120 minutes after infusion of levcromakalim or placebo
  Change in blood pressure (systolic and diastolic) measured in mmHg following infusion of levcromakalim compared to placebo in patients with migraine with aura

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thomsen AV, Al-Karagholi MA, Hougaard A, Ostrowski SR, Ashina M. Effects of levcromakalim in patients with migraine aura without headache: An experimental study. Cephalalgia. 2024 Aug;44(8):3331024241274366. doi: 10.1177/03331024241274366. PMID 39161224
- [Derived] Thomsen AV, Al-Karagholi MA, Hougaard A, Ostrowski SR, Pedersen OB, Hansen TF, Ashina M. Investigations of the migraine-provoking effect of levcromakalim in patients with migraine with aura. Cephalalgia. 2024 Mar;44(3):3331024241237247. doi: 10.1177/03331024241237247. PMID 38501895